CLINICAL TRIAL: NCT06853132
Title: Baduanjin With Resistance Training Program for Elderly Patients With Osteoporosis and Lumbar Disc Herniation
Brief Title: Baduanjin With Resistance Training Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Yale-China Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000039398
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Osteoporosis; Lumbar Disc Herniation
MeSH Terms: conditions — Osteoporosis; Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: Patients with LDH and OP who will be treated and undergo surgery will be recruited as potential participants from two spinal wards at the Second Xiangya Hospital of Central South University (Class A hospital) in Changsha City, Hunan Province.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants will receive conventional (usual) treatment: continue with their original treatment, medication, and diet habits. After spinal surgery, two nurses trained according to this study protocol will teach participants standard guidance for lumbar and back exercises, which will include exercise suggestions and health education.
- BDJ with resistance training (Experimental): BDJ exercise combined with resistance training and conventional (usual) treatment in the experimental group. Two nurses will provide training to ensure that participants can perform the movements skillfully and coherently.
  Interventions: Behavioral: Baduanjin with Resistance Training Program

INTERVENTIONS:
Behavioral: Baduanjin with Resistance Training Program — Baduanjin with Resistance Training Program
  Arms: BDJ with resistance training

SUMMARY:
The purpose of this study is to improve symptoms of Lumbar Disc Herniation (LDH) and Osteoporosis (OP) by implementing an evidence-based Baduanjin exercise to reduce pain and increase muscle strength and quality of life in Chinese patients. This study will provide new sights of exercise of elderly patients with LDH and OP for elderly patients.

DETAILED DESCRIPTION:
Participants in the control group will continue with their conventional post surgery treatment as follows: comprehensive post-operative care and educational handouts that include guidelines for lumbar and back exercises to improve recovery and promote spinal health. In addition, participants will receive three interactive Q&A sessions before discharge (pre-operation, post-operation, and on the day of discharge). During these sessions, patients can discuss their concerns and ask questions about their recovery.

Participants in the experimental group will continue to receive their conventional post surgery treatment in addition to BDJ as follows: Individual session training (admission to week 1 post-surgery), no training week 2, Group session I (week 3 and 4), Group session 2 (week 5-12) and perform independent exercises during which participants will have to keep an exercise diary (week 13-24).

Data collection will be conducted through in-person visits at baseline and Week 1, followed by phone calls at Week 12 and Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with LDH and OP based on the chart and clinical diagnostic criteria.
* Age of female patients ≥ 45 years，age of male patients ≥ 50 years.
* Visual analogue scale (VAS) ≥ 3 points.
* Surgical operation will be performed during the 7-day admission period.
* Mandarin speakers.

Exclusion Criteria:

* Severe primary diseases: ulcerative colitis, gastrointestinal bleeding, pancreatitis, lung cancer, pneumonia, acute respiratory distress syndrome or psychosis, depression, anxiety or substance abuse, identified by diagnosis and interview.
* Current engagement in regular physical activity routines over the past 3 months: aerobic exercises for at least 30 minutes, at least 3 times per week.
* Taken drugs within 3 months before enrollment: bisphosphonates, glucocorticoids, calcitonin, anticonvulsant drugs, heparin, etc.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of life measured by the Oswestry Disability Index (ODI) | Weeks 0, 1, 12, and 24
  ODI is the most widely accepted scales for assessing quality of life and the severity of disability caused by back pain. It assesses the impact of back pain on various daily activities. The ODI is a questionnaire containing 10 items covering disability caused by low back pain. Each item is assessed on a six-level ordinal scale with "0" describing "no limitation" and "5" describing "extreme limitation or an inability to function", with higher values representing a greater extent of disability. The total score is converted to a percentage to determine the severity of disability. Scores are interpreted as follows: 0-20% (minimal disability), 21-40% (moderate disability), 41-60% (severe disability), 61-80% (crippled), and 81-100% (bed-bound or exaggerating symptoms). The Cronbach's alpha of this scale was 0.89.
Change in Muscle strength by the Five Times Sit-to-Stand Test (FTSS) | Weeks 0, 1, 12, and 24
  The researchers need to record the total time spent going from sit to stand. At last, the test will be performed three times, and the final average in seconds is taken. Each patient was given 2 minutes intervals for rest. The time it takes to complete the five times sit-to-stand test (FTSST) varies by age and gender. Healthy adults complete the test in ≤ 10 seconds; times ≥15 seconds indicate increased fall risk and mobility impairments. The Cronbach alpha 0.99, and the reliability was 0.97.
Change in physical activity level by the International Physical Activity Questionnaire (IPAQ). | Weeks 0, 1, 12, and 24
  The IPAQ-LC is a widely used tool for assessing physical activity levels in various populations. This scale requires participants to complete 31 questions across four activity domains (transportation, work, household, and leisure time), and includes sections on walking, moderate and vigorous activity, and sedentary behaviors (sitting and lying awake]. The exercises recorded must last at least 10 minutes each time. To calculate a total activity score, the reported activity is assigned a Metabolic Equivalents (MET) value based on its intensity.
  (1) Low Activity Level: <600 MET minutes/ a week; (2) Moderate Activity Level: 600~3000 MET minutes/ a week; (3) > 3000 MET minutes/ a week.
  The Cronbach's alpha of this scale was 0.88.

SECONDARY OUTCOMES:
Change in Exercise self-efficacy by the Self-Efficacy for Exercise Scale (SEE) | Weeks 0, 1, 12, and 24
  This scale is designed to test individual's confidence to exercise in the face of barriers to exercise. It consists of 9 items, with scores ranging from 0 to 10 representing the exercise confidence levels. A score of 0 indicates "no confidence", while a score of 10 indicates "very confident". Total score range is 0-90. Higher scores reflect a greater level of exercise self-efficacy. The Cronbach alpha for this scale is 0.93.
Change in exercise benefit by the Exercise Benefits and Barriers Scale (EBBS) | Weeks 0, 1, 12, and 24
  This scale assesses the perceived benefits and barriers to exercise among patients. The EBBS consists of 43 items that evaluate the perceived benefits of exercise and factors that hinder participation. It includes two dimensions: exercise benefits and exercise barriers. A 4-point Likert scale is used (1 = "strongly disagree", 4 = "strongly agree"). The total score ranges from 43 to 172, with higher scores indicating more positive perceptions of exercise benefits and fewer perceived barriers. The Cronbach alphas for the overall scale and the two subscales are 0.86, 0.95, and 0.86, respectively.
Incidence of complications after surgery | Week 1
  Complications will be recorded by registered nurses. The data will be collected by clinical chart reviews and patient interviews. The incidence of complication after surgery will be calculated by the number of new complications / total number of participants in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Soohyun Nam, PhD, APRN, ANP-BC, FAHA, FAAN, Principal Investigator — Yale University
Locations (1):
- Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No